CLINICAL TRIAL: NCT07092397
Title: Artificial Intelligence-based Tumor Microenvironment Analysis for Prognosis Prediction in Gallbladder Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JooKyung Park, Professor, Samsung Medical Center
Other Study IDs: SMC-2022-03-136
Record Dates: First submitted 2025-07-13; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Gallbladder Cancer
Keywords: gallbladder cancer
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study aims to investigate the prognostic significance of artificial intelligence (AI)-powered analysis of tumor-infiltrating lymphocytes (TILs) and the tumor microenvironment (TME) in patients with resected gallbladder cancer. Using hematoxylin and eosin (H&E)-stained slides, the study quantifies spatial TME features, including TIL density, tertiary lymphoid structures, and fibroblast density, to identify potential TME-related risk factors associated with survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent curative surgery for gallbladder cancer.

Exclusion Criteria:

* Patients who did not achieve R0 resection.
* Patients with metastatic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with gallbladder cancer who underwent curative-intent surgery with R0 resection at Samsung Medical Center between 2010 and 2020 formed the main study cohort. An external validation cohort included patients with gallbladder cancer at Asan Medical Center between 2017 and 2022 with available archived hematoxylin and eosin-stained slides for AI-powered tumor microenvironment analysis. Patients with inadequate tissue samples were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of surgery (or diagnosis) to the date of death from any cause or the last follow-up, assessed up to 165 months

SECONDARY OUTCOMES:
Disease-free survival | From date of surgery to the date of disease recurrence, assessed up to 165 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
There is no current plan to publicly share individual participant data (IPD). However, de-identified data may be shared upon reasonable request, subject to approval by the institutional review board and compliance with data protection regulations.